CLINICAL TRIAL: NCT00520572
Title: A Randomised, Double-Blind (With Open Comparator Etanercept Limb), Placebo-Controlled, Phase IIb, Multicentre Study to Evaluate the Efficacy of 4 Doses of AZD9056 Administered for 6 Months on the Signs and Symptoms of Rheumatoid Arthritis in Patients With Active Disease Receiving Background Methotrexate or Sulphasalazine
Brief Title: A 6-month Randomised, Double-blind, Open Arm Comparator, Phase IIb, With AZD9056, in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1520C00001
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AZD9056; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 1 (Active Comparator): Etanercept 50mg, subcutaneous, once weekly
  Interventions: Drug: Etanercept
- 2 (Experimental): 50mg oral, once daily
  Interventions: Drug: AZD9056
- 3 (Experimental): 100 mg oral, once daily
  Interventions: Drug: AZD9056
- 4 (Experimental): 200 mg oral, once daily
  Interventions: Drug: AZD9056
- 5 (Experimental): 400mg once, daily
  Interventions: Drug: AZD9056
- 6 (Placebo Comparator): oral, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9056
  Arms: 2; 3; 4; 5
Drug: Etanercept
  Arms: 1
Drug: Placebo
  Arms: 6

SUMMARY:
The purpose of this study is to confirm that AZD9056 is effective in treating rheumatoid arthritis with regard to signs and symptoms and to determine what dose is favourable over a 6-month treatment period. Patients will receive background treatment with either Methotrexate or Sulphasalazine

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA with active disease defined as: ≥4 swollen joints and ≥6 tender/painful joints, and either have (blood tests) elevated erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP). At least one of the following: documented history and current presence of positive rheumatoid factor (blood test), baseline radiographic erosion.

Be receiving either oral (tablets) or subcutaneous/intramuscular (injection) methotrexate for at least 6 months prior to randomisation.

Exclusion Criteria:

* Any other inflammatory disease in addition to RA that may interfere with the study (e.g. polymyalgia rheumatica, giant cell arteritis, reactive arthritis, e t c). Current chronic pain disorders including fibromyalgia and chronic fatigue syndromes. Persistently abnormal liver function enzymes (blood test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2007-08; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Keystone, MD, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL; Zoltan Koroknai, MD, D.E.A.A., Study Chair — Omnicare Clinical Research
Locations (51):
- United States (8):
  - Research Site, Aventura, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Petoskey, Michigan
  - Research Site, Syracuse, New York
  - Research Site, Portland, Oregon
  - Research Site, Olympia, Washington
- Argentina (5):
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Planta Baja San Juan
  - Research Site, San Miguel de Tucumán
- Australia (4):
  - Research Site, Woolloongabba, Queensland
  - Research Site, Woodsville, South Australia
  - Research Site, Victoria Park, Western Australia
  - Research Site, George Town
- Research Site, Hasselt, Belgium
- Canada (2):
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
- Czechia (3):
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- France (3):
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Tours
- Mexico (6):
  - Research Site, Cd. Juarez
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Tapachula
  - Research Site, Tijuana
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
- Romania (6):
  - Research Site, Brasov, Brașov County
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Ploieşti
  - Research Site, Sf. Gheorghe
- Research Site, Saint Petersburg, Russia
- Slovakia (3):
  - Research Site, Bansky Bystrica
  - Research Site, Bratislava
  - Research Site, Piešťany

REFERENCES:
- [Derived] Keystone EC, Wang MM, Layton M, Hollis S, McInnes IB; D1520C00001 Study Team. Clinical evaluation of the efficacy of the P2X7 purinergic receptor antagonist AZD9056 on the signs and symptoms of rheumatoid arthritis in patients with active disease despite treatment with methotrexate or sulphasalazine. Ann Rheum Dis. 2012 Oct;71(10):1630-5. doi: 10.1136/annrheumdis-2011-143578. PMID 22966146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled on 01 August 2007, the last participant completed the study on 08 April 2009. Participants were recruited from 59 centres in 12 countries in Australia, Canada, Europe, Russia, South America, and the USA.
Pre-assignment Details: Male/female participants with active rheumatoid arthritis (and on background methotrexate or sulphasalazine) were randomly assigned to receive AZD9056 at 50, 100, 200 or 400 mg once daily, placebo or etanercept. It was planned to randomise approximately 360 participants, 60 to the open-label etanercept arm and 300 to the AZD9056 or placebo arms
Groups:
- AZD9056 50 mg: AZD9056 50 mg, oral tablets, once daily, double blinded
- AZD9056 100 mg: AZD9056 100 mg, oral tablets, once daily, double blinded
- AZD9056 200 mg: AZD9056 200 mg, oral tablets, once daily, double blinded
- AZD9056 400 mg: AZD9056 400 mg, oral tablets, once daily, double blinded
- Placebo: Placebo to AZD9056, oral tablets, once daily, double blinded
- Etanercept: Etanercept 50 mg, subcutaneous injection, once weekly, open label
Period: Overall Study
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Started | 64 (Participants randomised. One of these participants did not subsequently receive treatment.) | 64 (Participants randomised.) | 64 (Participants randomised. One of these participants did not subsequently receive treatment.) | 64 (Participants randomised.) | 65 (Participants randomised.) | 64 (Participants randomised.)
Completed | 52 (Participants completed the study.) | 50 (Participants completed the study.) | 49 (Participants completed the study.) | 50 (Participants completed the study.) | 53 (Participants completed the study.) | 62 (Participants completed the study.)
Not Completed | 12 | 14 | 15 | 14 | 12 | 2
Not completed — Adverse Event | 9 | 3 | 6 | 9 | 7 | 2
Not completed — Withdrawal by Subject | 0 | 9 | 5 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Incorrect enrollment | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Oral corticotherapy for acute urticaria | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Long break in taking Medication | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did not receive Treatment | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept | Total
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64 | 383
Age Continuous [Mean (Standard Deviation); unit: Years] | 52 (12.8) | 54 (11.5) | 50 (11.9) | 52 (11.8) | 51 (11.9) | 51 (10.8) | 51.7 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 51 | 59 | 54 | 55 | 329
  Male | 7 | 10 | 12 | 5 | 11 | 9 | 54

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20 Response (ACR20) at 6 Months
Description: The number of participants with greater to or equal to 20% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 6 months' treatment
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64
Participants | 23 | 26 | 23 | 21 | 21 | 42

2. Secondary Outcome: American College of Rheumatology 50 Response (ACR50) at 6 Months
Description: The number of participants with greater to or equal to 50% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 6 months' treatment.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64
Participants | 13 | 8 | 9 | 13 | 11 | 30

3. Secondary Outcome: American College of Rheumatology 70 Response (ACR70) at 6 Months
Description: The number of participants with greater to or equal to 70% improvement in the ACR composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, disease activity and physical function; physician's assessment of disease activity; and CRP) after 6 months' treatment
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64
Participants | 6 | 7 | 5 | 5 | 3 | 15

4. Secondary Outcome: Disease Activity Score (Based on 28 Joint Count) (DAS28) at 6 Months.
Description: Change from baseline in the DAS28 composite score (a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of disease activity; and ESR) after 6 months' treatment. A change of zero indicates no effect of treatment and a negative change of 1.2 indicates a clinically important improvement in symptoms. (The DAS scale runs from 0 to 10, with the higher scores indicating worse RA symptoms).
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64
Composite score | -1.2 (1.27) | -1.4 (1.63) | -1.1 (1.47) | -1.4 (1.37) | -1 (1.24) | -2.3 (1.38)

5. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) at 6 Months.
Description: Change from baseline in HAQ-DI (a measure of patients assessment of physical function scored between zero and 3) after 6 months' treatment, calculated as score at 6 months minus score at baseline. A change of zero indicates no effect of treatment and a negative change of 0.22 or greater indicates an improvement in symptoms. (The HAQ-DI scale runs from 0 to 3, with higher scores indicating greater disability).
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Number analyzed (Participants) | 63 | 64 | 63 | 64 | 65 | 64
Composite score | -0.3 (0.57) | -0.3 (0.51) | -0.2 (0.5) | -0.3 (0.55) | -0.3 (0.46) | -0.6 (0.66)

ADVERSE EVENTS:
Arm/Group | AZD9056 50 mg | AZD9056 100 mg | AZD9056 200 mg | AZD9056 400 mg | Placebo | Etanercept
Serious Adverse Events (participants affected / at risk) | 2/63 | 0/64 | 1/63 | 1/64 | 1/65 | 2/64
Other Adverse Events (participants affected / at risk) | 17/63 | 24/64 | 20/63 | 29/64 | 20/65 | 11/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AZD9056 50 mg (N=63) | AZD9056 100 mg (N=64) | AZD9056 200 mg (N=63) | AZD9056 400 mg (N=64) | Placebo (N=65) | Etanercept (N=64)
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0/37 | 0
Non-Cardiac Chest Pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ureteral Polyp (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9056 50 mg (N=63) | AZD9056 100 mg (N=64) | AZD9056 200 mg (N=63) | AZD9056 400 mg (N=64) | Placebo (N=65) | Etanercept (N=64)
Nausea (Gastrointestinal disorders) | 3 | 7 | 2 | 7 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 5 | 7 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4 | 6 | 3 | 0
Bronchitis (Infections and infestations) | 3 | 4 | 0 | 2 | 2 | 1
Rheumatoid Atheritis (Musculoskeletal and connective tissue disorders) | 8 | 6 | 4 | 6 | 12 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 3 | 1 | 2
Headache (Nervous system disorders) | 3 | 3 | 7 | 10 | 4 | 0
Hypertension (Vascular disorders) | 2 | 4 | 2 | 3 | 0 | 6

LIMITATIONS AND CAVEATS:
Hybrid ACR, ACRn, individual ACR components, Erythrocyte sedimentation rate, Short-form-36, Rheumatoid Arthritis Quality of Life, Patient Assessment of Fatigue and DEXA X-ray scanning did not provide extra information so are not presented

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less